CLINICAL TRIAL: NCT06213363
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase Ib/II Clinical Study to Evaluate the Efficacy, Safety and Pharmacokinetics of TCR1672 Tablets in Patients With Refractory Chronic Cough
Brief Title: A Phase Ib/II Clinical Study in Patients With Refractory Chronic Cough
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCR1672-II-01
Record Dates: First submitted 2023-12-15; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-12

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCR1672 tablet (Experimental): TCR1672 tablet
  Interventions: Drug: TCR1672 tablet
- TCR1672 placebo (Placebo Comparator): TCR1672 placebo
  Interventions: Drug: TCR1672 tablet

INTERVENTIONS:
Drug: TCR1672 tablet — All potential participants proceed to the screening period (7-14 days) after voluntarily signing the informed consent form, and the investigators conduct eligibility assessment for the participants as per the inclusion and exclusion criteria. 72patients with RCC are planned to be enrolled in this study. All participants will firstly be randomized at a ratio of 1:1:1 to receive one of the three oral doses of three times a day TCR1672 (20mg, 40mg, 60mg). Then patients will further be randomized to two treatment sequences, Dosing Sequence 1 and Dosing Sequence 2. Participants in Dosing Sequence 1 will be given TCR1672 Tablets for 1 weeks, followed by a 1-week washout period, and then crossover to 1-week placebo treatment. Participants in Dosing Sequence 2 will be firstly administered 1-week placebo treatment, followed by a 1-week washout period, and then crossover to TCR1672 tablets for 1-week treatment.

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled Phase Ib/II clinical trial to evaluate the effectiveness, safety, tolerability and pharmacokinetics (PK) of TCR1672 Tablets in patients with refractory chronic cough.

DETAILED DESCRIPTION:
All potential participants proceed to the screening period (7-14 days) after voluntarily signing the informed consent form, and the investigators conduct eligibility assessment for the participants as per the inclusion and exclusion criteria. 72patients with RCC are planned to be enrolled in this study. All participants will firstly be randomized at a ratio of 1:1:1 to receive one of the three oral doses of three times a day TCR1672 (20mg, 40mg, 60mg). Then patients will further be randomized to two treatment sequences, Dosing Sequence 1 and Dosing Sequence 2. Participants in Dosing Sequence 1 will be given TCR1672 Tablets for 1 weeks, followed by a 1-week washout period, and then crossover to 1-week placebo treatment. Participants in Dosing Sequence 2 will be firstly administered 1-week placebo treatment, followed by a 1-week washout period, and then crossover to TCR1672 tablets for 1-week treatment. TCR1672 Tablets will be administered orally after meal. No dose adjustments are allowed during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants who can understand and are willing to complete this trial in strict accordance with the clinical trial protocol, and voluntarily sign the informed consent form;
2. Age ≥ 18 years (subject to the age specified in the valid document at the time of signing the informed consent form);
3. Male participants weighing ≥ 50 kg and female participants weighing ≥ 45 kg, and BMI < 35kg/m2;
4. History of chronic cough for more than 1 year, and definitely diagnosed as refractory chronic cough or chronic cough of unknown cause. See Appendix 2 for the diagnostic criteria;
5. Chest imaging within 5 years prior to screening and after the onset of chronic cough did not show abnormal changes that in the opinion of the investigator may contribute to the chronic cough;
6. The 100-mm cough Visual Analogue Scale (VAS) score ≥ 40 mm at screening and baseline;
7. The cough recorder at screening showed an average of 10 or more coughs per hour while awake;
8. Participants of childbearing potential and their sexual partners are willing to take one or more effective non-drug contraceptive measures and have no plans to donate sperm or ova from the time of screening until 6 months after the last dose of study drug; Female participants should be non-pregnant and non-lactating, and should meet at least 1 of the following conditions:

   1. Not a woman of childbearing potential (WOCBP) as defined in the appendix;
   2. Is a WOCBP and agrees to follow the contraception requirements in the appendix for the duration of the study and for at least 6 months after the last dose of the study;
   3. The WOCBP has a negative blood pregnancy test prior to the first dose of study drug;
   4. If the blood pregnancy result is positive, the participant must be withdrawn from the study;
   5. Refer to the Study Flow Chart for additional pregnancy testing requirements during and after the study;
   6. Investigators are responsible for reviewing medical and menstrual history to see whether the requirements for highly effective contraception will be met so as to reduce the risk of including females with early undetected pregnancy.

Exclusion Criteria:

1. Pre-bronchodilator forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) < 70% of the expected value at screening;
2. History of upper or lower respiratory tract infection (including bacterial, fungal, viral and other pathogenic microorganism infections) or recent significant change in pulmonary conditions (including acute exacerbation of respiratory disease or significant change in chest imaging) within 4 weeks prior to screening or randomization;
3. Diagnosed as chronic obstructive pulmonary disease (COPD), bronchiectasis, idiopathic pulmonary fibrosis (IPF), active pulmonary tuberculosis before screening;
4. Past medical history of hypogeusia or taste disorder, or known taste abnormality;
5. With malignancy within 5 years prior to screening (except adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ);
6. Moderate renal insufficiency: glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 prior to screening or prior to randomization;
7. Moderate to severe hepatic insufficiency (Child-Pugh Class B or C) prior to screening or prior to randomization;
8. History of unstable or worsening cardiovascular disease prior to screening or prior to randomization, including but not limited to: unstable angina, myocardial infarction, thromboembolism;
9. Those who are smoking or have quitted smoking for less than 1 year, or have a smoking history of annual consumption of more than 20 pack-years at screening;
10. Recent (within the past 1 year) history of drug or alcohol abuse or dependence;
11. Known hypersensitivity to any ingredient of this medication;
12. Systemic or topical use of drugs or foods that may affect the PK characteristics of the study drug, including strong inducers, strong inhibitors or substrates of CYP2C19 and CYP3A, and drinking grapefruit or grapefruit juice within 14 days prior to screening and during the trial (see Table 6 for details);
13. Systemic or topical use of antitussive drugs, including opioids, pregabalin, gabapentin, dextromethorphan, traditional Chinese medicine and over-the-counter drugs with antitussive effect, etc., within 4 weeks prior to screening and during the trial [participants are allowed to receive a stable (≥ 4 weeks prior to the first dose of study drug) treatment for cough etiology, including antihistamines, leukotriene receptor antagonists, inhaled or oral glucocorticoids, long-acting bronchodilators, etc., or receive stable (≥ 8 weeks prior to the first dose of study drug) treatment with proton pump inhibitors];
14. Receiving an angiotensin converting enzyme inhibitor currently or within 3 months prior to screening;
15. Participation in any other clinical study with the last dose of an study drug within 4 weeks prior to screening, or within 5 half-lives at screening (whichever is longer);
16. Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg at screening and baseline (the test should be performed after resting for at least 5 minutes and the criterion is still met after a repeat examination);
17. Family history of long QT syndrome and sudden death, or significant ECG abnormalities at screening, including but not limited to: QTcF interval > 450 ms, atrial fibrillation or flutter, heart rate < 40 beats/min or > 110 beats/min, second or third degree atrioventricular block, left bundle branch block;
18. Clinically significant abnormalities in laboratory test results at screening, including but not limited to:

    1. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) or glutamyl transpeptidase (GGT) > 2 times the upper limit of normal, and total bilirubin > 1.5 times the upper limit of normal;
    2. Creatinine > times the upper limit of normal;
    3. Coagulation abnormalities including but not limited to abnormal platelet count (< 100 × 103/mm3), prolonged PT or INR ≥ 1.5;
19. Positive hepatitis B virus surface antigen, or positive hepatitis B virus core antibody, negative hepatitis B virus surface antibody and positive HBV-DNA, or positive hepatitis C virus antibody or positive HCV-RNA, or positive treponema pallidum antibody, or positive human immunodeficiency virus (HIV) antibody at screening;
20. Pregnant or breast-feeding;
21. Any past or current acute or chronic illness, psychiatric illness, or laboratory abnormality that, in the judgment of the investigator, may compromise the safety or compliance of the participant, or affect the absorption of the study drug and study assessments, or render the participant unable to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy Endpoint | 1 week
  Change from baseline in 24-hour cough frequency after 1-week treatment
Safety Endpoints | 4 week
  Severity and incidence of treatment emergent adverse events (TEAEs) from the first dose to the end of follow-up

IPD SHARING:
Plan to Share IPD: No